CLINICAL TRIAL: NCT05526261
Title: Benign Thyroid Nodules / Benign Goiter. What Subjective Problems Are Improved With an Operation and Can This be Predicted Preoperatively?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ervin Beka, General Surgeon MD, Linkoeping University
Other Study IDs: 2020-00022
Record Dates: First submitted 2022-08-16; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hemithyroidectoy — Hemithyroidectomy it is a surgical procedure where half of the thyroid gland is operated.

SUMMARY:
Nodules in the thyroid gland are common. Patients discover these lumps either because of their visible size increase or because of local discomforts such as difficulty swallowing, difficulty breathing or voice changes. The thyroid gland is in close connection with the esophagus, trachea and the vocal nerve. Thus, a lump in the thyroid gland can cause pressure symptoms from these organs. In the event of such complaints, patients are referred for investigation. If it turns out that the patient has a lump in the thyroid gland ("goiter"), further investigation is carried out with an ultrasound examination and sampling with a needle from the lump (puncture).

At present, most thyroid nodules are examined cytologically, ie the thyroid nodules are punctured with a thin needle and the cells that are obtained are analyzed by a cytologist. The material is graded according to Bethesda classification. Higher grading is associated with a higher risk that the tuber is malignant. Lower grading is associated with a lower probability that the tuber can be malignant. If these patients are operated on, it is usually with the hope that their local ailments improve.

We want to investigate which patients who have a lump in the thyroid gland and experience pressure problems experience an improvement after a thyroid operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a thyroid nodule who have local problems and where surgery (hemithyroidectomy) is planned
* 18 years or older
* Bethesda I-IV

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patientens with compression symptoms in the neck
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement | One year follow upp
  Which sypmtoms become better after hemithyroidectomy

SECONDARY OUTCOMES:
Comparision of questionnaries | 2024
  The patients are going to fill in 4 different questionnaries in 3 different time intervalls. Before the operation, 1 month and 1 year efter the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Gimm, Professor, Study Director — Professor Oliver Gimm
Locations (1):
- Linköpings University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No